CLINICAL TRIAL: NCT02780180
Title: A Randomized, Double-blind, Multi-centre Study to Assess Safety and Efficacy of Incremental Doses of QGC001 in Patients With NYHA Class II/III Chronic Heart Failure (HF) With Left Ventricular Systolic Dysfunction Versus Placebo.
Brief Title: QUantum Genomics Incremental Dosing in Heart Failure - QUID-HF
Acronym: QUID-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QUID-HF_v5.0_20171120
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Aminopeptidase A inhibitor; Heart Failure; Up-titration; Dose-Response Relationship, Drug; Pharmacokinetics; Patient Safety; Treatment Efficacy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QGC001 (Experimental): QGC001 from 50mg to 500mg capsule twice daily, for 28 days, oral use
  Interventions: Drug: QGC001
- Placebo (Placebo Comparator): Placebo, capsule twice daily, for 28 days, oral use
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGC001
  Arms: QGC001
Drug: Placebo — Lactose capsule manufactured to mimic QGC001 50 mg and 250 mg
  Arms: Placebo

SUMMARY:
Heart Failure (HF) a common clinical condition characterized by either by a heart that does not pump sufficiently or becomes stiff. A variety of mechanisms contribute to progressive cardiac remodeling and dysfunction.

A new therapeutic approaches by preventing activation of the brain neuromodulatory pathway, may lead to improve HF.

QCG001 is a prodrug of EC33, a aminopeptidase A (APA) inhibitor. QCG001 has been shown to be an antihypertensive agent in animal models.

This study investigates the safety and efficacy of QGC001 in HF patients.

DETAILED DESCRIPTION:
Despite advances in care, prognosis remains poor once overt Heart Failure (HF) has developed. HF is a common clinical condition characterized by either by a heart that does not pump sufficiently or becomes stiff and it is associates with higher incidences of patient illness and death in both case. A variety of mechanisms contribute to progressive cardiac remodeling and dysfunction.

A new therapeutic approaches by preventing activation of the brain neuromodulatory pathway, may lead to improve HF.

QCG001 is a prodrug of EC33, a specific and selective of the aminopeptidase A (APA) inhibitor. QCG001 has been shown to be an antihypertensive agent in animal models.

This study investigates the safety and efficacy of QGC001 up-titrated form 50mg twice daily to a maximum of 500 mg twice daily, on patients with worsening chronic HF during 28 days and 7 days after discontinuation (day 35).

6 European countries are involved in this study (France, Netherlands, Germany, Norway, Poland and United Kingdom) including 20 investigational hospitals. Patients would be followed during 35 days and inclusion period lasts until December 2017.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form prior to any study procedure
* Adult male subjects and female subjects without childbearing potential.
* Clinical diagnosis of CHF with history of NYHA class II-III for at least 3 months before randomisation.
* Documented left ventricular ejection fraction (LVEF) < 40% measured by any modality within the previous 12 months in the subject's medical history.
* Subjects must also have at least one local measurement of BNP level ≥ 300 pg/mL or NT-proBNP level ≥ 1200 pg/mL (preferred assay, local laboratory) at the screening visit (maximum 7 days before randomisation).
* eGFR > 30 mL/min/1.73 m2 (MDRD) at screening.
* Serum potassium < 5.0 mmol/L at screening.
* Systolic blood pressure < 110 mmHg (average of 3 consecutive measurements) at screening.
* Prescribed to optimal pharmacologic therapy per "ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2016", or based on the updated current clinical practice, unless contra-indicated or not-tolerated, and on a stable dose for at least 30 days prior to enrolment (the dosage of the drugs cannot be increased or decreased respectively by more than double or half of initial dosage).
* Taking oral loop diuretics at doses < 250 mg furosemide daily (or equivalent).

Exclusion Criteria:

* BMI > 45 kg.m-2.
* Patients who require the use of HF IV therapy or oral furosemide > 250 mg (or equivalent) at any time during the 48 hours immediately before randomisation.
* Patients with unstable angina, myocardial infarction, PTCA, coronary artery bypass graft, cerebral vascular accident, or transient ischemic attack within previous 3 months (90 days) before enrolment.
* Patients whose primary cause of heart failure is mitral or aortic valve disease or congenital heart disease or hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis) or myocarditis.
* Patients with "new" permanent atrial fibrillation (AF), discovered within 3 months prior to randomization.
* Heart rate > 110 beats/min at screening.
* Patients scheduled for Pacemaker (including ICD, CRT), Angioplasty, CABG or LVAD within the next 3 months.
* Patients with severe documented chronic obstructive lung disease (COPD), defined as chronic need for oxygen therapy
* eGFR < 30 mL/min/1.73 m2 (MDRD) at screening.
* Decrease in eGFR greater than 20% within 3 weeks prior to the screening visit.
* Serum potassium > 5.0 mmol/L at screening.
* Systolic blood pressure < 110 mmHg or with signs or symptoms of hypotension.
* Symptomatic hypotension or orthostatic hypotension defined by a decrease of systolic blood pressure of more than 30 mm Hg in the standing vs. sitting position at screening and at the basal SBP of the D0 (before having taken the study medication).
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstrated of a QTc interval > 450 ms) AND QRS < 100 ms. In case of QRS enlargement > 100 ms (i-e bundle branch block, pacemakers) QT does not accurately reflect repolarization and may not be calculated.
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g. hypokalemia, family history of long QT Syndrome).
* The use of concomitant medications that prolong the QT/QTc interval.
* Insulin-requiring diabetic patients (including type 1 Diabetes).
* History of angioneurotic edema.
* Severe liver failure at screening defined by a value of ALAT and/or ASAT≥ 5 from the normal value.
* Patients involved in any interventional clinical study, patients enrolled in Registries and/or in non-interventional studies may participate.
* Patients who take an investigational or non-approved treatment.
* Women of childbearing potential.
* Patients with a prior cardiac transplant or patients currently on the list for cardiac transplantation.
* Patient with hypersensitivity to the active substance or to one of the other components of the trial preparation.
* Patients in whom an allergy requiring chronic treatment is known or exists.
* Patients with a history of previous illnesses of neurological or psychiatric nature that affect the Central Nervous System.
* Patients with a life expectancy of less than 12 months per physician judgment.
* Frail patient who, in the opinion of the investigator will not be able to follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Relative decrease in NT-proBNP | 28 days
  Percentage of subjects with a relative decrease in NT-proBNP of more than 30% from Baseline to day 28.
Blood pressure change | 28 days
  Blood pressure changes at each visit (D7, D14, D21, D28), compared to the Baseline measure

SECONDARY OUTCOMES:
Blood biochemistry | 35 days
  blood biochemistry at D7, D14, D21, D28 and D35.
Urinary biochemistry | 35 days
  electrolytes, urinary osmolarity at D7, D14, D21, D28 and D35.
Change of NT-proBNP | 35 days
  Changes in central lab values of NT-proBNP at D7, D14, D21, D28 and D35.
Change of BNP | 35 days
  Changes in central lab values of BNP at D7, D14, D21, D28 and D35.
Change of selected biomarker levels | 28 days
  Changes in central lab values from baseline in selected biomarker levels (biomarkers involved in the pathophysiology of the disease, which will be decided later) at Day 7, Day 14, Day 21, Day 28
Quality of life Minnesota Living with Heart Failure Score | 28 days
  Quality of life Minnesota Living with Heart Failure Score and D0 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Faiez Zannad, MD, Principal Investigator — Centre d'investigation clinique CHU-Nancy
Locations (23):
- Czechia (2):
  - Hospital of Fridek-Mistek P.O., Frýdek-Místek
  - General University Hospital, Prague
- France (9):
  - Hôpital Louis Pradel, Bron
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHRU Nancy, Nancy
  - Hôpital Laennec, Nantes
  - Hôpital Pitié Salpêtrière, Paris
  - Georges Pompidou European Hospital, Paris
  - hôpital Charles Nicolle, Rouen
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Charity Universitatsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Klinik für Innere Medizin III, Homburg
- Hungary (2):
  - Heart and Vascular Center of Semmelweis University, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Centre, Maastricht
- Stavanger University Hospital, Stavanger, Norway
- Poland (2):
  - NZOZ ALL-MED Centrum Medyczne, Lodz
  - Clinical Military Hospital, Wroclaw
- United Kingdom (2):
  - University of Birmingham Institute of Cardiovascular Sciences City Hospital,, Birmingham, England
  - Ninewells Hospital, Dundee

IPD SHARING:
Plan to Share IPD: No
Individual participant date would be available only by the center via eCRF